CLINICAL TRIAL: NCT02688634
Title: The Role of Antibiotic Prophylaxis in Cleft Palate and Velopharyngeal Insufficiency Repair
Acronym: Cleft Palate
Status: Withdrawn | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500667
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Cleft Palate
Keywords: Cleft Palate Surgery; Antibiotic treatment
MeSH Terms: conditions — Cleft Palate | interventions — Amoxicillin; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment: Participants in this group are randomize to receive post-operative antibiotic of Amoxicillin x7 days, 20mg/kg orally every 6 hours to a maximum of 1.8g/day for a 7-day period. They will be evaluated for infection, fistula formation, and dehiscence upon discharge and at 30-day follow-up based on standards of care.
  Interventions: Drug: Amoxicillin
- Non-Treatment: Participants in this group will be randomize to no post-operative antibiotic. They will be evaluated for infection, fistula formation, and dehiscence upon discharge and at 30-day follow-up based on standards of care.

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin will be given as: 7 days, 20mg/kg orally every 6 hours to a maximum of 1.8g/day for a 7-day period.
  Other Names: Antibiotics
  Groups: Treatment

SUMMARY:
Cleft Lip and Palate surgical repair is one of the most common procedures performed by Plastic and Reconstructive Surgeons in the World. With this in mind, it is curious that no consensus exists regarding the usage of postoperative antibiotics or the effects this might have on wound complications such as cellulitis, dehiscence, or fistula formation. The surgical bed in cleft lip/palate repair is known to harbor a myriad of pathological organisms, indeed the human bite is one of the more clinically and microbiologically significant injuries to treat. This research study is to elucidate the role, if any, that prophylactic antibiotics have in the prevention of complications post cleft palate (CP) and VPI repair and potentially establish a new paradigm of care.

DETAILED DESCRIPTION:
This will be a randomized prospective research study. Participants who will undergo an elective CP or VPI surgery will be randomized to receive either 1) antibiotics or 2) nothing postoperatively. All participants will be evaluated for infection, fistula formation, and dehiscence upon discharge and at 30-day follow-up based on standards of care.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 1 month to 60 years
2. Subjects undergoing independently scheduled elective Cleft Palate of VPI repair
3. Do not meet any exclusion criteria

Exclusion Criteria:

1. Any repeat repair
2. Symptoms of upper respiratory infection
3. Immunosuppressed
4. Allergy to Amoxicillin or any other Penicillins
5. Antibiotic usage <2weeks prior to scheduled surgery other than immediate pre-operative antibiotics
6. Inability to follow up

Ages: 1 Month to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects undergoing independently scheduled elective Cleft Palate of VPI repair at an area hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Infection rates between the groups | 30 days
  Analysis of infection is based on a 7 point scale to allow for broadened data but can be evaluated in a binary fashion for ≥ 4 indicating infection and <4 as no infection. A χ2 test and Fisher's exact test for p<0.05 will be used to determine significance of the difference in complication (cellulitis and upper respiratory infection) rates between the two groups.
Dehiscence and fistula formation between the groups | 30 days
  Both dehiscence and fistula formation will also be recorded as a binary present/not present data point to determine the significance of the difference in complication rates between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Lentz, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health at Shands Hospital, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No